CLINICAL TRIAL: NCT00079222
Title: Randomized Trial Of Safety And Tolerability Of Intravenous/Oral Voriconazole Versus Intravenous/Oral Itraconazole For Long-Term Antifungal Prophylaxis In Allogeneic Hematopoietic Stem Cell Transplant Recipients
Brief Title: Voriconazole Compared With Itraconazole in Preventing Fungal Infections in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Mary Territo, University of California, Los Angeles
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000355116; UCLA-0307071
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2013-01

CONDITIONS: Cancer
Keywords: infection; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated childhood acute lymphoblastic leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; accelerated phase chronic myelogenous leukemia; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative disease, unclassifiable; previously treated myelodysplastic syndromes; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory hairy cell leukemia; refractory multiple myeloma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; recurrent ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; poor prognosis metastatic gestational trophoblastic tumor; disseminated neuroblastoma; recurrent neuroblastoma; recurrent ovarian germ cell tumor; previously treated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma; recurrent Wilms tumor and other childhood kidney tumors; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; juvenile myelomonocytic leukemia; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Infections; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Myeloproliferative Disorders; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Multiple Myeloma; Leukemia, Hairy Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Recurrence; Mycosis Fungoides; Sezary Syndrome; Testicular Neoplasms; Carcinoma, Ovarian Epithelial; Neuroblastoma; Wilms Tumor; Breast Neoplasms; Leukemia, Myelomonocytic, Juvenile; Lymphoma, B-Cell, Marginal Zone; Congenital Abnormalities | interventions — Itraconazole; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: itraconazole
Drug: voriconazole

SUMMARY:
RATIONALE: Antifungals, such as voriconazole and itraconazole, may be effective in preventing fungal infections in patients who are undergoing allogeneic stem cell transplantation.

PURPOSE: This randomized clinical trial is studying voriconazole to see how well it works compared to itraconazole in preventing fungal infections in patients who are undergoing allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the safety and tolerability of voriconazole vs itraconazole for the prevention of fungal infections in patients undergoing allogeneic hematopoietic stem cell transplantation.

OUTLINE: This is a randomized study. Patients are stratified according to donor type (related vs unrelated). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning after allogeneic hematopoietic stem cell transplantation (AHSCT), patients receive voriconazole IV twice daily on days 1-14 and then orally* twice daily on days 15-100.
* Arm II: Beginning after AHSCT, patients receive itraconazole IV twice daily on days 1-2, once daily on days 3-14, and then orally* twice daily on days 15-100.

NOTE: *Patients unable to tolerate oral medication may continue IV medication beyond day 14.

In both arms, treatment continues in the absence of unacceptable toxicity or an invasive fungal infection. Patients requiring corticosteroid therapy for graft-versus-host disease continue to receive voriconazole or itraconazole beyond day 100.

Patients are followed until day 180 post-transplantation.

PROJECTED ACCRUAL: A total of 150 patients (75 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing allogeneic hematopoietic stem cell transplantation
* No invasive yeast infection within the past 8 weeks

  * Colonized or superficial infection allowed
* No documented or probable aspergillus or mold infection within the past 8 weeks
* Patients with a history of candidemia must have negative blood cultures and no clinical signs of candidemia

PATIENT CHARACTERISTICS:

Age

* 12 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior allergy or intolerance to imidazoles or azoles (e.g., fluconazole, itraconazole, voriconazole, ketoconazole, miconazole, or clotrimazole)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 1 week since prior amphotericin B or fluconazole for candidemia
* No concurrent therapy with any of the following:

  * Rifampin
  * Rifabutin
  * Phenobarbital
  * Phenytoin
  * Carbamazepine
  * Oral midazolam
  * Triazolam
  * Terfenadine
  * Astemizole
* Concurrent topical antifungal agents for superficial fungal infections allowed

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-11; Primary Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary C. Territo, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States